CLINICAL TRIAL: NCT06875037
Title: Patient-reported Outcomes of Accelerated Upper Canine Retraction With Low-amperage Electrical Stimulation: A Randomized Controlled Trial
Brief Title: Patient-related Outcomes When Accelerating Upper Canine Retraction With Fixed Orthodontic Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-4-2025
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Stimulation Group (Experimental): Patients in this group will undergo conventional orthodontic treatment combined with electrical stimulation for the retraction of upper canines.
  Interventions: Device: Electric stimulation removable appliance
- Conventional Traction Group (Active Comparator): Patients in this group will receive conventional orthodontic treatment without any acceleration method.
  Interventions: Procedure: Traditional orthodontic fixed appliance without accleration

INTERVENTIONS:
Device: Electric stimulation removable appliance — The device will be used with the fixed appliance to accelerate orthodontic tooth movement (i.e., canine retraction).
  Arms: Electrical Stimulation Group
Procedure: Traditional orthodontic fixed appliance without accleration — The traditional method of canine retraction will be employed using fixed appliances. No additional appliances will be used to activate orthodontic tooth movement.
  Arms: Conventional Traction Group

SUMMARY:
Patients will be screened in the Orthodontics Department of the Faculty of Dentistry, Damascus University, and those who meet the inclusion criteria will be included. Then, the initial diagnostic records (diagnostic plaster casts, intra- and extra-oral photographs, and radiographs) will be studied to ensure the selection criteria are accurately met.

This study aims to compare two groups of patients with Class II malocclusion. Experimental Group: Patients in this group will undergo maxillary canine retraction using the traditional sliding technique with fixed appliances, supplemented by electrical current stimulation.

Control Group: Patients in this group will undergo maxillary canine retraction using the traditional sliding technique with fixed appliances, without any acceleration method.

DETAILED DESCRIPTION:
Maxillary canine retraction can be lengthy, and various methods have been employed to accelerate it. Electrical current stimulation has shown promise as a technique for speeding up tooth movement. However, only a limited number of studies have been documented in the literature. Controlled clinical studies are necessary to evaluate the effectiveness of this procedure in accelerating tooth movement, its impact on pain responses, and other patient-centred outcomes.

Participants will be selected from patients attending the Orthodontics Department at the Faculty of Dentistry, Damascus University. Eligible patients with Class II/Division I malocclusion who meet the inclusion criteria will be invited to participate in this trial after being screened by the researcher. Informed consent will be obtained from all patients who agree to join the study after receiving an information sheet.

Alignment and leveling will be performed using pre-adjusted fixed orthodontic appliances consisting of 0.022 x 0.028-inch metal brackets with the MBT prescription. The traditional wiring sequence will be followed until a 0.019 x 0.025-inch stainless steel base wire is in place.

Maxillary first premolars will be extracted during the leveling and alignment phase, with more than two months between the completion of the alignment phase and the extraction. This ensures that the phenomenon of regional acceleration generated by the extraction does not affect the rate of tooth movement.

Canine retraction will be achieved using closed-coil nickel-titanium (NiTi) springs extending from the upper first molar band hook to the canine bracket hook. A force of 150 grams will be applied to each side, and the force will be checked using a force meter at each appointment (every two weeks) until the canine retraction is complete, achieving a Class I canine relationship.

A small electrical current will be applied to the upper maxillary canine area using a removable intraoral appliance containing a micro electrical circuit. Each patient in the experimental group will be asked to wear the electrical accelerator in their mouth for 5 hours daily.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 17 to 28 years.
* Class II Division 1 malocclusion (according to Angle's classification) requires the extraction of the upper first premolar as part of the orthodontic treatment plan.
* Mild to moderate skeletal Class II (ANB = 5-7).
* Overjet of 5 to 10 mm.
* Normal or vertical growth patterns (MM ≥ 26; SN-MP ≥ 33; Y Axis ≥ 65)

Exclusion Criteria:

* Moderate to severe dental crowding.
* Missing teeth in the upper arch.
* Previous orthodontic treatment.
* Health conditions or long-term medication.
* Periodontal disease.
* Poor oral hygiene.
* Smoking

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in the perception of pain | Questionnaires will be completed at the following assessment times: on the 1st, 3rd, and 7th days of the first, second, and third months from the start of the canine retraction.
  Patients will be asked to rate their pain perception with the question, "What is the degree of pain you are experiencing at this moment?" They will indicate their pain level by placing a mark on a horizontal 100-mm line. The left end of the line represents no pain (VAS=0), and the right end signifies maximum (unimaginable) pain (VAS=100).
Change in the perception of discomfort | Questionnaires will be completed at the following assessment times: on the 1st, 3rd, and 7th days of the first, second, and third months from the start of the canine retraction.
  Patients will be asked to rate their perception of discomfort with the question, "What is the degree of discomfort you are experiencing at this moment?" They will indicate their level of discomfort by placing a mark on a horizontal 100-mm line. The left end of the line represents no discomfort (VAS=0), while the right end signifies maximum (unimaginable) discomfort (VAS=100).

SECONDARY OUTCOMES:
Change in difficulty swallowing | Questionnaires will be completed at the following assessment times: on the 1st, 3rd, and 7th days of the first, second, and third months from the start of the canine retraction.
  Patients will be asked to rate their perception of difficulty swallowing with the question, "What is the degree of difficulty swallowing you are experiencing at this moment?" They will indicate their level of difficulty swallowing by placing a mark on a horizontal 100-mm line. The left end of the line represents no difficulty swallowing (VAS=0), while the right end signifies maximum difficulty swallowing (VAS=100).
Change in the chewing ability | Questionnaires will be completed at the following assessment times: on the 1st, 3rd, and 7th days of the first, second, and third months from the start of the canine retraction.
  Patients will be asked to rate their perception of chewing ability with the question, "What is the degree of difficulty you are experiencing in chewing?" They will indicate their level of chewing difficulty by placing a mark on a horizontal 100-mm line. The left end of the line represents no difficulty (VAS=0), while the right end signifies maximum difficulty in mastication (VAS=100).
Change in the speech ability | Questionnaires will be completed at the following assessment times: on the 1st, 3rd, and 7th days of the first, second, and third months from the start of the canine retraction.
  Patients will be asked to rate their perception of speech ability with the question, "What is the degree of difficulty you are experiencing in speech?" They will indicate their level of speech difficulty by placing a mark on a horizontal 100-mm line. The left end of the line represents no difficulty (VAS=0), while the right end signifies maximum difficulty (VAS=100).
Change in analgesic consumption | Questionnaires will be completed at the following assessment times: on the 1st, 3rd, and 7th days of the first, second, and third months from the start of the canine retraction.
  Patients will be asked the following question about "Analgesic Consumption": "Did you need to take pain analgesics?" Analgesic consumption is assessed by inquiring if the study participant took analgesics, using a two-point scale (1. Yes or 2. No).
Patients' satisfaction | Questionnaires will be filled at the end of the fourth month of the canine retraction
  Patients will be asked to evaluate their satisfaction with orthodontic treatment with the question, "How satisfied are you with your orthodontic treatment?" Satisfaction for both groups will be assessed by having the study participant place a mark on a horizontal 100-mm line to indicate their level of satisfaction. The left end of the line represents no satisfaction (VAS=0), while the right end signifies maximum satisfaction (VAS=100).
Recommendation of the procedure to a friend | Questionnaires will be filled at the end of the fourth month of the canine retraction
  Patients will be asked the following question about the likelihood of recommending the procedure to their friends: "Would you recommend this treatment to a friend?" Those in the experimental group will indicate their response using a two-point scale (1. Yes, or 2. No).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad N. Kheshfeh, DDS, Principal Investigator — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria; Mohammad Y. Hajeer, DDS MSc PhD, Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mousa MM, Hajeer MY, Burhan AS, Darwich KMA, Almahdi WH, Aljabban O, Awawdeh MA, Almasri IA. Patient-Reported Outcome Measures of Flapless Corticotomy with Low-Level Laser Therapy in En Masse Retraction of Upper Anterior Teeth: A Three-Arm Randomized Controlled Trial. Clin Pract. 2023 Nov 22;13(6):1501-1519. doi: 10.3390/clinpract13060132. PMID 38131681
- [Background] Mousa MM, Hajeer MY, Burhan AS, Almahdi WH. Evaluation of patient-reported outcome measures (PROMs) during surgically-assisted acceleration of orthodontic treatment: a systematic review and meta-analysis. Eur J Orthod. 2022 Dec 1;44(6):622-635. doi: 10.1093/ejo/cjac038. PMID 35796046
- [Background] Shaadouh RI, Hajeer MY, Mahmoud GA, Almasri IA, Jaber ST, Alam MK. Patient-reported outcomes during accelerating the en-masse retraction of the upper anterior teeth using low-intensity electrical stimulation: a randomized controlled trial. Prog Orthod. 2024 May 13;25(1):17. doi: 10.1186/s40510-024-00517-3. PMID 38735912
- [Background] Alfailany DT, Hajeer MY, Awawdeh MA, Khursheed Alam M, Darwich KMA, Aljabban O, Latifeh Y, Alhaffar JB, Almasri IA. Evaluation of Patient-Reported Outcome Measures (PROMs) Associated With the Acceleration of Canine Retraction by Piezosurgery in Comparison With Low-Level Laser Therapy: A Three-Arm Randomized Controlled Clinical Trial. Cureus. 2024 Jan 7;16(1):e51779. doi: 10.7759/cureus.51779. eCollection 2024 Jan. PMID 38192530
- [Background] Charavet C, Lecloux G, Jackers N, Maes N, Lambert F. Patient-reported outcomes measures (PROMs) following a piezocision-assisted versus conventional orthodontic treatments: a randomized controlled trial in adults. Clin Oral Investig. 2019 Dec;23(12):4355-4363. doi: 10.1007/s00784-019-02887-z. Epub 2019 Apr 6. PMID 30955096
- [Derived] Kheshfeh MN, Hajeer MY, Alam MK, Al Hinnawi MF, Latifeh Y. Patient-reported outcome measures of accelerated upper canine retraction with low-amperage electrical stimulation: A randomized controlled trial. Int Orthod. 2025 Oct 3;24(1):101077. doi: 10.1016/j.ortho.2025.101077. Online ahead of print. PMID 41045595